CLINICAL TRIAL: NCT03575923
Title: Evaluating the Impact of Improvements in Urban Green Space on Older Adults' Physical Activity and Wellbeing: a Natural Experimental Study
Acronym: GHIA
Status: Completed | Type: Observational
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Jack Benton, Principal Investigator, University of Manchester
Other Study IDs: NE/N013530/1
Record Dates: First submitted 2018-06-11; First posted 2018-07-03 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Physical Activity and Wellbeing
Keywords: Physical activity; Wellbeing; Urban green space; Older adults; Natural experiment; Protocol; GHIA
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (12):
- Intervention site 1: 2 planted trees; bulb planting
  Interventions: Behavioral: Urban street greening
- Comparison site 1A
- Comparison site 1B
- Intervention site 2: 12 planted trees; bulb planting; artificial tree decorations (string lights)
  Interventions: Behavioral: Urban street greening
- Comparison site 2A
- Comparison site 2B
- Intervention site 3: 3 planted trees; artificial tree decorations (string lights, tree socks)
  Interventions: Behavioral: Urban street greening
- Comparison site 3A
- Comparison site 3B
- Intervention site 4: 8 planted trees; bulb planting; artificial tree decorations (string lights, tree socks)
  Interventions: Behavioral: Urban street greening
- Comparison site 4A
- Comparison site 4B

INTERVENTIONS:
Behavioral: Urban street greening — The interventions are located on four publicly accessible sites; the total size of the floor area of green space in each of the intervention sites is small, ranging from 0.09 to 0.35 acres. Components of the interventions include tree and flower planting (expected to bloom by March 2018) and artificial tree decorations such as strings of small electric lights and tree socks (the interventions are hereafter collectively referred to as urban street greening). The total cost for all components across all four intervention sites is approximately £6,000, although this excludes artist fees connected to the project. All components of the interventions were implemented within a one week period in November 2017 by two arborists, two local artists, staff members at Southway Housing Trust, and local community members from Old Moat and a local school.
  Groups: Intervention site 1; Intervention site 2; Intervention site 3; Intervention site 4

SUMMARY:
Background: Creating or improving urban green space has the potential to be an effective and sustainable way to increase physical activity and improve other aspects of wellbeing in older adults. However, the size and quality of the existing evidence base is weak. There is particularly a lack of studies on older adults and in the United Kingdom. This study aims to evaluate the effect of four small local street greening intervention projects on older adults' physical activity and wellbeing over a one-year period. The street greening includes tree and flower planting, and artificial tree decorations. These projects are based in a deprived urban neighbourhood in Greater Manchester, United Kingdom.

Methods: Eight unimproved comparison sites were selected to compare with the intervention sites. The researchers will measure physical activity and two other behavioural indicators of wellbeing (Connect: connecting with other people; and Take Notice: taking notice of the environment) using a newly developed observation tool. It is thought that the largest effect of the interventions will be on Take Notice behaviour due to improvements in the aesthetic quality of green space at the intervention sites. Baseline data collection occurred in September 2017 before the interventions were installed in November 2017. Follow-up data collection will be repeated in February/ March 2018 (6 months) and September 2018 (12 months).

Discussion: The present study offers a rare opportunity to evaluate the before-and-after effects of small-scale changes in urban green space, in an understudied population (older adults) and setting (United Kingdom). Although the interventions are expected to have small effects on peoples' behaviour, this study will address key weaknesses in previous studies.

ELIGIBILITY:
Inclusion Criteria:

° All individuals (infants, children, teens, adults, older adults) entering the target area during observation periods

Exclusion Criteria:

° Any individuals that request their data to be removed from the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study is focused on older adults and therefore primary analyses will only consider data from older adults. Secondary analyses will consider data from adults.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2017-09-04 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Take Notice behaviour | 12 months
  The primary outcome will be a count per observation period of Take Notice behaviour at 12 months. Take Notice behaviour is the primary outcome because the interventions are expected to improve the aesthetic quality of green space by providing visual information of value to users, thus causing more overt appreciation in the intervention sites.

SECONDARY OUTCOMES:
Take Notice behaviour | 6 months
  The investigators will also assess a count per observation period of Take Notice behaviour at 6 months.
Overall count of older adults | 6 months
  The secondary outcome will be the overall count of older adults per observation period.
Overall count of older adults | 12 months
  The secondary outcome will be the overall count of older adults per observation period.

OTHER OUTCOMES:
Sedentary behaviour | 6 months
  Additional exploratory analyses will assess a count per observation period separately for each physical activity level (Sedentary, Walking, Vigorous) and Connect behaviour.
Sedentary behaviour | 12 months
  Additional exploratory analyses will assess a count per observation period separately for each physical activity level (Sedentary, Walking, Vigorous) and Connect behaviour.
Walking behaviour | 6 months
  Additional exploratory analyses will assess a count per observation period separately for each physical activity level (Sedentary, Walking, Vigorous) and Connect behaviour.
Walking behaviour | 12 months
  Additional exploratory analyses will assess a count per observation period separately for each physical activity level (Sedentary, Walking, Vigorous) and Connect behaviour.
Vigorous physical activity | 6 months
  Additional exploratory analyses will assess a count per observation period separately for each physical activity level (Sedentary, Walking, Vigorous) and Connect behaviour.
Vigorous physical activity | 12 months
  Additional exploratory analyses will assess a count per observation period separately for each physical activity level (Sedentary, Walking, Vigorous) and Connect behaviour.
Connect behaviour | 6 months
  Additional exploratory analyses will assess a count per observation period separately for each physical activity level (Sedentary, Walking, Vigorous) and Connect behaviour.
Connect behaviour | 12 months
  Additional exploratory analyses will assess a count per observation period separately for each physical activity level (Sedentary, Walking, Vigorous) and Connect behaviour.

CONTACTS AND LOCATIONS:
Locations (1):
- Greater Manchester, Multiple Locations, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There are no individual participant data

REFERENCES:
- [Derived] Benton JS, Anderson J, Cotterill S, Dennis M, Lindley SJ, French DP. Evaluating the impact of improvements in urban green space on older adults' physical activity and wellbeing: protocol for a natural experimental study. BMC Public Health. 2018 Jul 27;18(1):923. doi: 10.1186/s12889-018-5812-z. PMID 30053861